CLINICAL TRIAL: NCT03538171
Title: A Randomized Phase III Clinical Study of Entinostat/Placebo in Combination With Exemestane in Chinese Patients With Hormone Receptor-positive Advanced Breast Cancer
Brief Title: Ph3 Study of Exemestane With or Without Entinostat in Chinese Patients With Hormone Receptor-Positive, Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taizhou EOC Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EOC103A3101
Record Dates: First submitted 2018-04-27; First posted 2018-05-29 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — entinostat; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM Entinostat+Exemestane (Active Comparator): Patients receive Exemestane orally (PO) once daily (QD) on days 1-28 and Entinostat PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entinostat; Drug: Exemestane
- ARM Placebo+Exemestane (Placebo Comparator): Patients receive Exemestane as in Arm A and placebo PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo; Drug: Exemestane

INTERVENTIONS:
Drug: Entinostat — Entinostat will be repeatedly administered PO on days 1, 8, 15 and 22 of each treatment cycle. Exemestane PO once daily on day 1-28.
  Arms: ARM Entinostat+Exemestane
Drug: Placebo — Patients receive Exemestane as in Arm A and placebo PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Arms: ARM Placebo+Exemestane
Drug: Exemestane — Exemestane PO once daily on day 1-28.

SUMMARY:
The purpose of this randomized phase III trial is to evaluate the clinical benefit of combining entinostat with exemestane in Chinese patients with HR-positive, HER2-negative, locally advanced or metastatic breast cancer, who have disease progression on endocrine therapy. Additionally，the safety, tolerability, and PK profile of the treatment combination are evaluated.

DETAILED DESCRIPTION:
This randomized phase III trial studies entinostat combination with exemestane to see how well they work compared to exemestane alone in treating Chinese patients with hormone receptor-positive, locally advanced or metastatic breast cancers.

Estrogen can drive the growth of breast cancer cells. Exemestane may fight breast cancer by lowering the amount of estrogen the body makes from tissue aromatase. Entinostat may enhance the anti-tumor effect of exemestane in breast cancer by helping to overcome tumor resistance via epigenetic modifications. Previous Phase II trial in US breast cancer patients have demonstrated significant effects of combined therapy in slowing disease progression and on patient survival when compared to exemestane alone. It is not yet known whether exemestane is more effective when combined with entinostat in Chinese patients with advanced breast cancer. In this parallel, randomized, double blind, active controlled study, we will study the effect of entinostat/placebo in combination with exemestane in Chinese patients with hormone receptor-positive, HER2 receptor-negative, locally advance or metastatic breast cancer, who have experienced disease progression with prior endocrine therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Female, age≥18 years and ≤75 years (For the Open-label study， only the patients with natural menopause or surgical ovariectomy are enrolled).

   Note: surgical ovariectomy is defined as bilateral oophorectomy.
3. The ECOG score is 0-1.
4. Life expectancy duration ≥12 weeks.
5. Estrogen receptor (ER) and/or progesterone receptor (PR) positive, human epidermal growth factor receptor 2 (HER-2) negative.

   1. ER and PR status should be histologically confirmed with staining of ≥ 1% cells.
   2. Positive human epidermal growth factor receptor 2 (HER-2) should be defined as positive ISH test or immunohistochemical test +++ or ++ with positive ISH amplification test.
   3. Receptor status may be based on any time during treatment prior to study randomization, and from any site (i.e. primary, recurrent, or metastatic).
6. The patient must have measurable or non-measurable but can only be bone metastasis Stage III /locally advanced or metastatic breast cancer (in accordance with the general evaluation criteria, RECIST Version 1.1). Bone metastasis includes osteolytic or mixed type (osteolytic and osteogenic).

   For Part 2 the Randomized, double-blind study: the ratio of patients with non-measurable lesion (only bone metastasis) should be ≤ 20%; not required for Part 1-the Open-label study.

   Notes:
   1. Evaluation of lesions must be performed within 4 weeks prior to the randomization. The radiological examination includes cranial MRI (magnetic resonance imaging), thoracic and abdominal contrast-enhanced CT (computed tomography, the lower limit of abdominal scan must reach anterior superior iliac spine). MRI is optional in patients who are allergic to the contrast substance. It needs to ensure that the lesions should be scanned and evaluated in accordance with the requirement in the general evaluation criteria RECIST version 1.1.
   2. Non-measurable lesion is defined as all the other lesions, including small foci (the maximum diameter<10 mm or minor axis of pathological lymph node ≥10 mm but <15 mm) and unmeasurable foci (meningeal foci, ascites, hydrothorax, pericardial effusion, pelvic effusion, inflammatory breast cancer, carcinomatous lymphangitis of skin or lung, abdominal mass that can't be diagnosed or followed up by radiology, and cystic lesion).
7. At least one previous treatment of endocrine therapy other than Exemestane.
8. As previous adjuvant therapy,Exemestane is allowed to be used, if the disease-free interval is >12 months after discontinuation of Exemestane.
9. For the patients with metastatic breast cancer who have already received at most one chemotherapeutic regimen，the end of chemotherapy should be at least 4 weeks before the randomization.
10. The end of previous radiotherapy should be at least 2 weeks before the randomization, and the patient must have recovered from the toxicity of radiotherapy (grade 1 or below).
11. The patient is allowed to receive the medications to regulatebone metabolism, for example, bisphosphonates and RANK-L (nuclear factor κB ligand receptor activator, e.g., denosumab); the bone metabolism-regulating therapy needs to be initiated 1 week prior to the first administration of treatment in the clinical trial, the same drug must be used throughout the clinical trial, except that actual clinical situation that requires amendment to the therapeutic regimen;
12. Patients must have adequate hematological, hepatic and renal function one week (7 days) prior to the Run-in period in open-label study and prior to randomization in randomized, double-blind study, which are defined as below:

    1. Haemoglobin (Hgb) ≥ 90 g/L;
    2. platelet count ≥ 100×109/L
    3. Absolute neutrophil count ≥ 1.5×109/L
    4. Serum creatinine ≤ 2.0 mg/dL
    5. Total bilirubin < 1.5 ×ULN (upper limit of normal) (≤3 mg/dL in case of Gilbert syndrome);
    6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; ALT and AST ≤5×ULN for liver metastasis.
13. Open-label study only enroll the patients with natural menopause or surgical ovariectomy. Postmenopausal, premenopausal/perimenopausal and menopausal female patients can be enrolled in the randomized, double-blind study; patients with childbearing potential must agree to use recognized effective methods for contraception (including condom containing sperm inactivation, vaginal septum, oral or injectable contraceptives, etc.) or abstain from sex life during participation in the study and within three months after discontinuation of the treatment.

Postmenopause is defined as:

1. Underwent irreversible surgical sterilization such as amputation of uterus, bilateral oophorectomy, but not tubal ligation;
2. Age≥60 years;
3. Age<60 years, natural menopause≥12 months, blood follicle stimulating hormone (FSH) and estradiol (E2) levels within the postmenopausal range (FSH>40 IU/L and E2<30 pg/mL) in case of no use of chemotherapy, Tamoxifen, Toremifene or ovariectomy in recent one year;
4. Age <60 years, currently using Tamoxifen or Toremifene, blood follicle stimulating hormone (FSH) and estradiol (E2) levels within the postmenopausal range (FSH>40 IU/L and E2<30 pg/mL).

Notes:

1. It will be considered as the premenopausal or perimenopausal state if the above criteria on menopause are not met;
2. The premenopausal/perimenopausal female patients can be enrolled only when they agree to use the concomitant drug LHRH agonist Goserelin, and need to start the dose of LHRH agonist at least 4 weeks prior to randomization;
3. If the patient has received other LHRH agonist prior to entry in the study, he/she must switch to Goserelin during the study.

Exclusion Criteria:

1. Previous or current metastatic foci in central nervous system, or leptomeningeal disease;

   Patients with stable symptoms of CNS metastasis can be accepted only during the open label phase, but the following conditions need to be met at the same time:

   The patient has lesions outside the CNS system. The CNS metastases did not involve the midbrain, pons, medulla oblongata or spinal cord.

   The patients did not receive whole brain radiotherapy within 6 weeks.

   - Confirmed that CNS disease remained stable for at least four weeks (including radiotherapy and/or surgical resection).

   Patients do not need hormone therapy for CNS diseases, such as dexamethasone combined with mannitol; Patients are unlikely to have any medical symptoms associated with CNS metastasis, such as headache, dizziness, nausea, vomiting, and intracranial hypertension.
2. Current or previous history of other malignant tumor (except for cured basal cell carcinoma or squamous cell carcinoma of skin, carcinoma in situ of cervix), unless taking radical therapy and no evidence of recurrence or metastasis in recent 5 years;
3. Uncontrolled or serious cardiovascular disease, for example, refractory angina pectoris, congestive heart failure within half a year prior to the screening; myocardial infarction within 12 months prior to screening; any history of clinically significant ventricular arrhythmia, prolonged QT interval; history of cerebrovascular accident, symptomatic coronary heart disease requiring drug therapy;
4. The 3rd space effusion (e.g., hydrothorax and ascites) which can not be controlled with drainage or other therapeutic method;
5. Patients with a history of immune deficiency, including HIV-positive;
6. Clinically significant abnormality in gastrointestinal function that may affect intake, transportation or absorption of oral administration of drugs (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
7. Unrecovered toxicity resulted from previous medication or toxicity, evaluation score is still > grade 1 (except alopecia);
8. Use of HDAC inhibitor (e.g., valproic acid, Entinostat, Vorinostat, chidamide, etc.) prior to enrollment or intended use of HDAC inhibitor during the study;
9. Known allergic to Exemestane, Entinostat or other drugs containing benzamide structure (e.g., Tiapride, Remoxipride, clebopride, etc.); allergic to Goserelin in premenopausal/perimenopausal female patients;
10. Any cognitive disorder resulted from mental or neurological disease, including epilepsy and dementia;
11. Clinically uncontrolled active infection, for example, acute pneumonia, active phase of hepatitis B (positive Hepatitis B surface antigen, and copy of DNA > upper limit of normal) two weeks (14 days) prior to the dose in the Open-label study and prior to randomization in the double-blind study;
12. Major surgery (judged by investigators in accordance with the previous history), major trauma or fracture 4 weeks (28 days) prior to the first dose in the Open-label study and prior to randomization in the double-blind study;
13. Organ transplant recipient;
14. Women who are pregnant or breastfeeding;
15. Patients who plan to receive other anticancer therapy or other investigational product during the study;
16. Participation in any other drug clinical trial 4 weeks (28 days) prior to the screening or currently receiving treatment in other clinical trials (except those who are participating in the follow-up of overall survival in one study);
17. Patients who are considered by investigators as inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
PFS (The Randomized Double-blinded Part) | From the day of randomization, assessment will be made every 8 weeks (±3 days) to the earliest of documented disease progression (PD) or death caused by any reason (whichever happens first), assessed up to 40 months.
  Progression Free Survival, defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). The distribution of PFS will be estimated using the Kaplan- Meier method, with 95% confidence intervals calculated using Greenwood's formula. In the primary analysis of PFS, differences in treatment effect will be tested using stratified log rank tests, stratifying on the randomization stratification factors. Stratified univariate and multivariable Cox proportional-hazard models will be built to estimate the hazard ratios (HRs) for treatment effect for PFS as a supportive analysis. In all analyses, P-values will be two-sided.

SECONDARY OUTCOMES:
OS (both the Open-label and Randomized Double-blinded parts) | From the day of first administration to the date of death from any cause, assessed up to 48 months.
  Overall Survival
Safety and tolerability (both the Open-label and Randomized Double-blinded parts) | From the first administration of the investigational product to 30 days after the last administration. The Randomized Double-blinded: assessed up to 48 months
  Incidence of toxicity graded according to National Cancer Institute CTCAE version 4.0. All treatment-emergent, baseline adverse events and hematological/biochemical toxicities based on laboratory measurements, as well as drug related AEs, will be summarized by both groups. The incidence of deaths and treatment-emergent serious AEs (defined as number of patients experiencing the AE divided by all treated patients) will be summarized and compared between Arm Entinostat+Exemestane and Arm Placebo+Exemestane. Also, the incidence of adverse events leading to discontinuation of investigational product and/or patient's withdrawal from the study will be summarized and listed.
ORR (both the Open-label and Randomized Double-blinded parts) | From the first administration on Day 1 Run-in Period or randomization day, evaluation will be made every 8 weeks (±3 days), until the earliest of documented PD or death caused by any reason (whichever happens first), assessed up to 48 months.
  Objective Response Rate, defined as the proportion of patients with complete response (CR) or partial response (PR) among all patients assessed per RESIST v1.1. Objective response in the two arms will be evaluated by comparing objective response rate (ORR, PR+CR) on the intention-to-treat patients with one-sided type I error of 2.5%. ORR will be summarized along with the exact binomial 95% confidence interval. In all analyses, P-values will be two-sided.
Pharmacokinetics (The Randomized Double-blinded Part) | Cycle 1 Day 1, within 3h and 5h after the administration; Cycle 1 Day 15,1h after the administration; Cycle 2 Day 1, within 72h prior to administration.
  Time at which maximum plasma concentration was observed.
CBR (both the Open-label and Randomized Double-blinded parts) | Estimated per 8 weeks (±3 days) from the first administration of the investigational product on Day 1 Run-in Period or randomization day, to the earliest of documented PD or death caused by any reason (whichever happens first),assessed up to 48 months.
  Clinical Benefit Rate, defined as CR+PR+SD≥ 24 weeks

OTHER OUTCOMES:
PBMC acetylation | Cycle 1 Day 1, prior to administration; ; Cycle 2 Day 1, prior to administration.
  To evaluate whether the efficacy of exemestane with entinostat varies with changes in acetylation status in peripheral blood mononuclear cells (PBMCs).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu B, Zhang Q, Hu X, Li Q, Sun T, Li W, Ouyang Q, Wang J, Tong Z, Yan M, Li H, Zeng X, Shan C, Wang X, Yan X, Zhang J, Zhang Y, Wang J, Zhang L, Lin Y, Feng J, Chen Q, Huang J, Zhang L, Yang L, Tian Y, Shang H. Entinostat, a class I selective histone deacetylase inhibitor, plus exemestane for Chinese patients with hormone receptor-positive advanced breast cancer: A multicenter, randomized, double-blind, placebo-controlled, phase 3 trial. Acta Pharm Sin B. 2023 May;13(5):2250-2258. doi: 10.1016/j.apsb.2023.02.001. Epub 2023 Feb 9. PMID 37250148